CLINICAL TRIAL: NCT06700616
Title: A Multicenter, Prospective Cohort Study in Patients With Myasthenia Gravis in China
Brief Title: A Study in Patients With Myasthenia Gravis in China
Acronym: MG Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9030R00001
Record Dates: First submitted 2024-09-30; First posted 2024-11-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Generalized Myasthenia Gravis; Refractory Myasthenia Gravis; Prospective Study; Observational Study; Cohort Study; Patient Registry; Chinese
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-center, prospective cohort study designed to characterize current clinical practice, clinical and patient-reported outcomes (PROs), disease prognosis, treatment patterns and healthcare resource utilization for Chinese patients with myasthenia gravis (MG). This study will enroll patients with MG as diagnosed by physician. Approximately 1,200 MG patients are intended to be recruited from approximately 40 sites across majority of regions in China. The clinical and PROs included MGFA class, MGFA PIS, MG-ADL (Activities of Daily Living), QMG (Quantitative MG score), MG QOL-15R, EQ-5D etc. All MG patients enrolled will be followed up every 6 months until end of 2027.

ELIGIBILITY:
Inclusion Criteria:

This study will enroll patients of all ages who are diagnosed with MG of all MGFA classifications by physicians.

1. Patients must have the following data to be enrolled in this study:

   * MGFA classification
   * MG-ADL score
2. MG patients or their legal guardians/representatives are able to sign the Informed Consent Form (ICF).

Exclusion Criteria:

1. Patients aged ≥18 years with ocular myasthenia gravis (MGFA class I) lasting for more than 2 years;
2. Patients who are currently participating in an interventional clinical trial cannot be enrolled in this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit patients diagnosed with MG by a physician. The diagnosis of MG patients newly diagnosed prior to enrollment should be based on the clinical characteristics of MG and at least one of the following criteria: (a) Positive serology tests for acetylcholine receptor antibody (AChR Ab), muscle-specific kinase antibody (MuSK Ab), or lipoprotein-related protein 4 (LRP4 Ab); (b) Results of electrophysiological studies (repetitive stimulation, single-fiber electromyography, or both) related to synaptic transmission disorder at the neuromuscular junction; (c) Positive pharmacological test results (such as neostigmine methylsulfate test). Previously diagnosed patients must have a documented MG diagnosis accepted by clinical physician.
Sampling Method: Non-Probability Sample
Enrollment: 1199 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | Every 6 months up to 3 years
  MGFA classification (e.g I, II, III, IV, V)
Treatment method | Every 6 months up to 3 years
  Targeted treatment methods (list of methods, including medication, immunoglobulin, plasma exchange, surgery etc. )
Patient-reported outcome | Every 6 months up to 3 years
  MG-Activities of Daily Living (MG-ADL, aggregated value in a scale, ranged 0- best to 24- worst)
Clinical outcome | Every 6 months up to 3 years
  MGFA Post-intervention Status (e.g. CSR, PR, MM)
Clinical outcome | Every 6 months up to 3 years
  Quantitative MG score (QMG, aggregated value in a scale, ranged 0- best to 39-worst)
Clinical outcome | Every 6 months up to 3 years
  Physician-reported MG crisis
Clinical outcome | Every 6 months up to 3 years
  Death
Patient-reported outcome | Every 6 months up to 3 years
  MG-Quality of Life 15-Revised (MG-QoL15-r, aggregated value in a scale for quality of life, ranged 0- best to 60- worst)
Patient-reported outcome | Every 6 months up to 3 years
  EuroQol-5D (separate value for five dimensions in a scale for quality of life)
Treatment duration | Every 6 months up to 3 years
  Therapies start and end date
Treatment dose | Every 6 months up to 3 years
  Dose (e.g. mg)
Treatment frequency | Every 6 months up to 3 years
  Frequency (e.g. times/day)

SECONDARY OUTCOMES:
Demographic factors | Baseline
  1. Age (years)
  2. Gender (male, female)
  3. Residence place (rural, urban)
  4. Education
  5. Household income
Healthcare resource utilization | Every 6 months up to 3 years
  MG-related hospitalization (days)
Cormobidity | Every 6 months up to 3 years
  Comorbidities (list of related diseases, e.g. autoimmune diseases, cardiovascular disease, hypertension, diabetes etc.)
Healthcare resource utilization | Every 6 months up to 3 years
  MG-related healthcare costs
MG diagnosis history | Every 6 months up to 3 years
  MG first time diagnosis date
Vital sign - blood pressure | Every 6 months up to 3 years
  Blood pressure (mmHg)
Laboratory test - blood cell test | Every 6 months up to 3 years
  Blood cell counts by cell type tests (e.g. counts/L)
Laboratory tests etc.) - MG-related antibodies | Every 6 months up to 3 years
  MG-related antibodies including AChR, MuSK, LRP4 etc. (positive or negative).
Vital sign - pulse | Every 6 months up to 3 years
  Pulse (count/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Fudong Shi, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (20):
- China (20):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Harbin
  - Research Site, Hebei
  - Research Site, Henan
  - Research Site, Inner Mongolia
  - Research Site, Jiangsu
  - Research Site, Lanzhou
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan

IPD SHARING:
Plan to Share IPD: Yes
Qualiﬁed researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identiﬁed individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home